CLINICAL TRIAL: NCT04741386
Title: The Immune-response and Safety of COVID-19 Vaccination in Patients With Chronic Kidney Disease, on Dialysis, or Living With a Kidney Transplant - A Prospective, Controlled, Multicenter Cohort Study by the RECOVAC Consortium
Brief Title: The REnal Patients COVID-19 VACcination Immune Response (RECOVAC IR) Study
Acronym: RECOVAC-IR
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Erasmus Medical Center (Other); Radboud University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, MD PhD, University Medical Center Groningen
Other Study IDs: NL76215.042.20
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Chronic Kidney Diseases
Keywords: SARS-CoV-2 vaccination; Antibody based immune response; SARS-CoV-2 specific T and B cell response
MeSH Terms: conditions — COVID-19; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — In total 3x50 ml heparin blood blood and 4x5 mL serum will be drawn and stored. In a subset of participants a total of 5 nasal strips will be collected and stored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort A: Patients with CKD stages 4 and 5
  Interventions: Biological: SARS-CoV-2 vaccination
- Cohort B: Patients on hemodialysis and peritoneal dialysis
  Interventions: Biological: SARS-CoV-2 vaccination
- Cohort C: Kidney Transplant Recipients
  Interventions: Biological: SARS-CoV-2 vaccination
- Cohort D: Controls
  Interventions: Biological: SARS-CoV-2 vaccination

INTERVENTIONS:
Biological: SARS-CoV-2 vaccination — All participants will receive two vaccinations against COVID-19 according to the manufacturer's instructions.

SUMMARY:
Rationale: COVID-19 is associated with severely increased morbidity and mortality in patients with severely impaired kidney function, on dialysis or alive with a kidney transplant. Therefore, effective SARS-CoV-2 vaccination would be of great clinical importance in these patients. However, SARS-CoV-2 vaccination studies have excluded patients with chronic kidney disease (CKD) so-far.

Objective: To assess the efficacy and safety of SARS-CoV-2 vaccination in patients with CKD stages 4/5, on dialysis or alive with a kidney transplant as compared to controls.

Study design: prospective, controlled multicenter study Study population: 175 patients with CKD stages 4/5 (eGFR < 30 ml/min/1.73m2), 175 on dialysis , 300 alive with a kidney transplant and 200 controls (partners or sibblings of patients) Intervention: SARS-CoV-2 vaccination according to standard of care. Blood will be drawn at 4 different time points (baseline and at day 28, month 6 and in a subset 28 days after a third vaccination).

Main study parameters/endpoints: The primary endpoint is the antibody based immune response on day 28 after the second vaccination. Participants will be classified as responders or non-responders based on a spike (S)1 specific antibody levels of >=10 or <10 BAU/mL. The percentage of responders of each patient cohort will be compared with the percentage responders in the control group. Safety is a secondary endpoint which will be reported in terms of percentage of solicited local and systemic adverse events (AEs)graded according to severity. Other secondary endpoints include longevity of the immune response at 6 months, antibody respons 28 days after a third vaccination and levels of SARS-CoV-2 specific T and B cell responses.

DETAILED DESCRIPTION:
OBJECTIVES

Primary objective:

To assess the antibody response after SARS-CoV-2 vaccination in patients with CKD stages 4/5, on dialysis or alive with a kidney transplant as compared to controls.

Secondary Objectives:

To assess in these groups of subjects after SARS-CoV 2 vaccination:

* durability of the antibody response
* the SARS-CoV-2-specific T and B cell response
* adverse events
* antibody response after third vaccination in patients on dialysis and kidney transplant recipients

Exploratory Objectives:

To assess in these groups of subjects after SARS-CoV 2 vaccination:

* the association between baseline (immune) parameters and the immune response to SARS-CoV-2 vaccination
* the neutralizing capacity of anti-COVID-19 antibodies
* the incidence of SARS-CoV-2 infection and outcome of COVID-19 disease during 6 months after SARS-CoV-2 vaccination and in a subset 28 days after third vaccination

STUDY DESIGN

This is a prospective, controlled multicenter cohort study to evaluate the efficacy and safety after SARS-CoV-2 vaccination in patients with CKD4/5, dialysis patients and kidney transplant recipients as compared to controls. Therefore, 4 cohorts will be included in this study.

* Cohort A: Patients with CKD stages 4 and 5 (eGFR <30 ml/min*1.73m2) (n = 175)
* Cohort B: Patients on hemodialysis and peritoneal dialysis (n = 175)
* Cohort C: Kidney Transplant Recipients (n= 300)
* Cohort D: Controls (n = 200)

Assessment of immune response:

Blood samples will be collected at baseline (i.e. prior to first vaccination) and 28 days, and 6 months after the second vaccination and in a subset 28 days after the third vaccination.

Evaluation other parameters:

To evaluate hematology parameters, liver and kidney function, additional blood samples will be collected at baseline, and 28 days and 6 months after the second vaccination.

Information on clinical course, incidence of SARS-CoV-2 infection, outcome of COVID-19 will be collected up to 6 months after second and in a subset 28 days after third vaccination for descriptive purposes.

METHODS

Main study parameter/endpoint:

The primary endpoint is the antibody based immune response to vaccination against COVID-19 on day 28 after the second vaccination as compared to controls.

Secondary study parameters/endpoints:

1. Duration and in-depth assessment of immune response through:

   * Measurement of SARS-CoV2 specific antibodies at 6 months after vaccination to test the durability of response
   * Assessment of SARS-CoV2 specific T and B cell response, 28 days, and 6 months after the second vaccination using a high throughput Interferon ɣ, IL-21 SARSCoV-2 specific T cell ELISPOT and SARS-CoV2 specific B cell memory ELISPOT.
2. Safety assessment through:

   - Incidence and severity of solicited AEs during 7 days after each vaccination
3. Antibody based immune response after third vaccination:

   * Measurement of SARS-CoV-2 specific antibodies at 28 days after third vaccination in patients on dialysis and kidney transplantation recipients.

Exploratory study parameters:

* Baseline (immune) parameters associated with vaccination response
* Neutralizing capacity of antibodies to test functionality
* In-depth flow-cytometric analyses for functional and phenotypical characterization of SARS-CoV-2 specific T cell responses will be performed followed by assessment of proliferative capacity, cytokine production and phenotypical markers in a subset of patients.
* Information on incidence of SARS-CoV-2 infection and outcome of COVID-19 disease during 6 months after second vaccination and in a subset 28 days after third vaccination will be collected.
* In a substudy in Radboudumc nasal strips will be collected and mucosal antibody response to COVID-19 analysed

ELIGIBILITY:
Inclusion Criteria:

1. All patients should be eligible for COVID-19 vaccination as described by the instructions of the manufacturer.
2. Age of 18 years or older
3. Capable of understanding the purpose and risks of the study, fully informed and given written informed consent
4. Either

   * CKD4/5, with an eGFR <30 ml/min*1.73m2 by CKD-EPI
   * Hemodialysis, or peritoneal dialysis
   * KT recipient at least 6 weeks after transplantation
   * Partner, sibling or family member of participating patient

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g. anaphylaxis) to any component of the study intervention(s)
* Multi-organ transplant recipients
* Previous or active COVID-19 disease
* Pregnancy or breastfeeding
* Active (haematological) malignancy
* Inherited immune deficiency
* Infection with Human Immunodeficiency Virus (HIV)
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.

Additional exclusion criterion for patients with CKD stages 4/5, on dialysis and controls:

- Individuals who receive maintenance treatment with immunosuppressive therapy in the 6 months before inclusion, including cytotoxic agents or systemic corticosteroids.

Additional exclusion criterion for controls:

- severely impaired kidney function, with an eGFR < 45 ml/min*1.73m2 by CKD-EPI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * At all four participating centers (UMCG, ErasmusMC, Radboudumc and Amsterdam UMC) out-patient clinics with at least 100 patients with CKD4/5 are available for recruitment in this study.
  * At all three participating centers approximately 50-100 hemodialysis and peritoneal dialysis patients are being treated, from this population eligible patients will be included.
  * Kidney transplant recipients at UMCG, Erasmus MC, Radboudumc and Amsterdam UMC will be eligible. In each participating center 130 to 200 patients receive a kidney transplant yearly, and per center 1000-2000 kidney transplant recipients are under regular outpatient follow-up.
  * Partners, siblings or family members of participating patients will be asked as controls.
Sampling Method: Non-Probability Sample
Enrollment: 854 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
The antibody based immune response to vaccination against COVID-19 as compared to controls | 28 days after the second vaccination
  Participants will be classified as responders or non-responders based on seroconversion with a threshold for seropositivity based on Receiver Operator Curve (ROC) analysis and set at 10 BAU/mL in individuals without measurable anti-S antibodies at baseline.

SECONDARY OUTCOMES:
Longevity of the antibody based immune response | 6 months after the second vaccination
  Decline in antibodies and change in antibody response (defined as an antibody concentration above or below 10 BAU/mL)
SARS-CoV2 specific T and B cell response | 28 days and 6 months after the second vaccination
  using a high throughput Interferon ɣ, IL-21 SARSCoV-2 specific T cell ELISPOT and SARS-CoV2 specific B cell memory ELISPOT
Incidence and severity of solicited adverse events | during 7 days after each vaccination
  Using questionaires
SARS CoV-2 spike-1 specific IgG antibody response after third COVID-19 vaccination | 28 days after the third vaccination
  5 drops of blood will be drawn by home finger-prick blood test in a subset of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Stephan F Sanders, MD PhD, Study Director — University Medical Center Groningen; Ron T Gansevoort, MD PhD, Principal Investigator — University Medical Center Groningen; Luuk B Hilbrands, MD PhD, Principal Investigator — Radboud University Medical Center; Marlies EJ Reinders, MD PhD, Principal Investigator — Erasmus Medical Center; Frederike J Bemelman, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Netherlands (4):
  - Radboud university medical center, Nijmegen, Gelderland
  - Amsterdam University Medical Center, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahn C, Amer H, Anglicheau D, Ascher NL, Baan CC, Battsetset G, Bat-Ireedui B, Berney T, Betjes MGH, Bichu S, Birn H, Brennan D, Bromberg J, Caillard S, Cannon RM, Cantarovich M, Chan A, Chen ZS, Chapman JR, Cole EH, Cross N, Durand F, Egawa H, Emond JC, Farrero M, Friend PJ, Geissler EK, Ha J, Haberal MA, Henderson ML, Hesselink DA, Humar A, Jassem W, Jeong JC, Kaplan B, Kee T, Kim SJ, Kumar D, Legendre CM, Man K, Moulin B, Muller E, Munkhbat R, Od-Erdene L, Perrin P, Rela M, Tanabe K, Tedesco Silva H, Tinckam KT, Tullius SG, Wong G. Global Transplantation COVID Report March 2020. Transplantation. 2020 Oct;104(10):1974-1983. doi: 10.1097/TP.0000000000003258. No abstract available. PMID 32243281
- [Background] Gansevoort RT, Hilbrands LB. CKD is a key risk factor for COVID-19 mortality. Nat Rev Nephrol. 2020 Dec;16(12):705-706. doi: 10.1038/s41581-020-00349-4. PMID 32848205
- [Background] Gezondheidsraad. Strategieën voor COVID-19-vaccinatie. Den Haag: Gezondheidsraad, 2020; publicatienr. 2020/23
- [Background] Hilbrands LB, Duivenvoorden R, Vart P, Franssen CFM, Hemmelder MH, Jager KJ, Kieneker LM, Noordzij M, Pena MJ, Vries H, Arroyo D, Covic A, Crespo M, Goffin E, Islam M, Massy ZA, Montero N, Oliveira JP, Roca Munoz A, Sanchez JE, Sridharan S, Winzeler R, Gansevoort RT; ERACODA Collaborators. COVID-19-related mortality in kidney transplant and dialysis patients: results of the ERACODA collaboration. Nephrol Dial Transplant. 2020 Nov 1;35(11):1973-1983. doi: 10.1093/ndt/gfaa261. PMID 33151337
- [Background] Hodgson SH, Mansatta K, Mallett G, Harris V, Emary KRW, Pollard AJ. What defines an efficacious COVID-19 vaccine? A review of the challenges assessing the clinical efficacy of vaccines against SARS-CoV-2. Lancet Infect Dis. 2021 Feb;21(2):e26-e35. doi: 10.1016/S1473-3099(20)30773-8. Epub 2020 Oct 27. PMID 33125914
- [Background] Katerinis I, Hadaya K, Duquesnoy R, Ferrari-Lacraz S, Meier S, van Delden C, Martin PY, Siegrist CA, Villard J. De novo anti-HLA antibody after pandemic H1N1 and seasonal influenza immunization in kidney transplant recipients. Am J Transplant. 2011 Aug;11(8):1727-33. doi: 10.1111/j.1600-6143.2011.03604.x. Epub 2011 Jun 14. PMID 21672157
- [Background] Kotton CN. Immunization after kidney transplantation-what is necessary and what is safe? Nat Rev Nephrol. 2014 Oct;10(10):555-62. doi: 10.1038/nrneph.2014.122. Epub 2014 Jul 29. PMID 25072119
- [Background] Mahase E. Covid-19: Vaccine candidate may be more than 90% effective, interim results indicate. BMJ. 2020 Nov 9;371:m4347. doi: 10.1136/bmj.m4347. No abstract available. PMID 33168562
- [Background] Reddy S, Chitturi C, Yee J. Vaccination in Chronic Kidney Disease. Adv Chronic Kidney Dis. 2019 Jan;26(1):72-78. doi: 10.1053/j.ackd.2018.10.002. PMID 30876620
- [Background] van Besouw NM, Yan L, de Kuiper R, Klepper M, Reijerkerk D, Dieterich M, Roelen DL, Claas FHJ, Clahsen-van Groningen MC, Hesselink DA, Baan CC. The Number of Donor-Specific IL-21 Producing Cells Before and After Transplantation Predicts Kidney Graft Rejection. Front Immunol. 2019 Apr 9;10:748. doi: 10.3389/fimmu.2019.00748. eCollection 2019. PMID 31024571
- [Background] Williamson EJ, Walker AJ, Bhaskaran K, Bacon S, Bates C, Morton CE, Curtis HJ, Mehrkar A, Evans D, Inglesby P, Cockburn J, McDonald HI, MacKenna B, Tomlinson L, Douglas IJ, Rentsch CT, Mathur R, Wong AYS, Grieve R, Harrison D, Forbes H, Schultze A, Croker R, Parry J, Hester F, Harper S, Perera R, Evans SJW, Smeeth L, Goldacre B. Factors associated with COVID-19-related death using OpenSAFELY. Nature. 2020 Aug;584(7821):430-436. doi: 10.1038/s41586-020-2521-4. Epub 2020 Jul 8. PMID 32640463
- [Derived] Vervoort JPM, Konijn WS, Jansen DEMC, Boersma C, de Zeeuw J, Ho-Dac-Pannekeet MM, Gansevoort RT, Messchendorp AL, Sanders JSF, de Wildt-Liesveld R. Patient engagement as a collaborative process in a large Dutch COVID-19 vaccination study (RECOVAC) - insight into the contribution of patient engagement and learnings for the future. Res Involv Engagem. 2024 Sep 13;10(1):96. doi: 10.1186/s40900-024-00622-x. PMID 39272117
- [Derived] Sanders JF, Messchendorp AL, de Vries RD, Baan CC, van Baarle D, van Binnendijk R, Diavatopoulos DA, Geers D, Schmitz KS, GeurtsvanKessel CH, den Hartog G, Kho MML, Koopmans MPG, van der Molen RG, Remmerswaal EBM, Rots N, Gansevoort RT, Bemelman FJ, Hilbrands LB, Reinders MEJ; VACcination Immune Response Study (RECOVAC) Collaborators. Antibody and T-Cell Responses 6 Months After Coronavirus Disease 2019 Messenger RNA-1273 Vaccination in Patients With Chronic Kidney Disease, on Dialysis, or Living With a Kidney Transplant. Clin Infect Dis. 2023 Feb 8;76(3):e188-e199. doi: 10.1093/cid/ciac557. PMID 35796536
- [Derived] Sanders JF, Bemelman FJ, Messchendorp AL, Baan CC, van Baarle D, van Binnendijk R, Diavatopoulos DA, Frolke SC, Geers D, GeurtsvanKessel CH, den Hartog G, van der Heiden M, Imhof C, Kho MML, Koopmans MPG, Malahe SRK, Mattheussens WB, van der Molen R, van Mourik D, Remmerswaal EBM, Rots N, Vart P, de Vries RD, Gansevoort RT, Hilbrands LB, Reinders MEJ; RECOVAC Collaborators. The RECOVAC Immune-response Study: The Immunogenicity, Tolerability, and Safety of COVID-19 Vaccination in Patients With Chronic Kidney Disease, on Dialysis, or Living With a Kidney Transplant. Transplantation. 2022 Apr 1;106(4):821-834. doi: 10.1097/TP.0000000000003983. PMID 34753894